CLINICAL TRIAL: NCT01262755
Title: Temple Registry for the Investigation of African American Gastrointestinal Disease Epidemiology
Acronym: TRIAGE
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Frank K. Friedenberg, Professor of Medicine, Temple University
Other Study IDs: K24DK083268 (NIH); K24DK083268 (NIH)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Gastroesophageal Reflux Disease; Functional Bowel Disorders
Keywords: GERD; IBS; Minority
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- African Americans: Consists of 450 African Americans living in the zip code surrounding Temple Hospital between the ages of 18 and 80.
  Interventions: Behavioral: Structured Interview

INTERVENTIONS:
Behavioral: Structured Interview — Subjects underwent a structured interview using a laptop computer and answered over 200 standardized questions. All patient had their height, weight, and waist circumference measured.

SUMMARY:
DESCRIPTION: Minimal data exists on the prevalence of gastroesophageal reflux disease in minority populations. Specific objectives of this K24 research project are to: (1) Provide an estimate of the prevalence of gastroesophageal reflux disease in an urban, African American population; (2) Determine whether specific risk factors including diet, tobacco use, physical activity, and psychosocial stress are important in the targeted population. We will also measure height, weight, and waist/hip circumference to determine the impact of central obesity on reflux. PUBLIC HEALTH RELEVANCE: This research will help doctors to understand the frequency and risks for esophageal reflux disease (heartburn) in African Americans.

DETAILED DESCRIPTION:
Treatment Plan

The goal of our survey will be to obtain responses from at least 450 self-described African Americans.

Method From our previous study we found that relying on responses from surveys placed in resident mailboxes (which need to be mailed back to us) is ineffective. For this study we have divided the zip code into roughly four equal quadrants using Broad Street and Erie Avenue as dividers. We will place a flyer in 1000 mail boxes in each quadrant by hand delivery. Hand delivery assures that mailings to vacated buildings will not occur. We hand delivered surveys in our previous study and encountered no problems. This will allow for a balanced representation from the entire zip code (see data collection section for further discussion of this point). The flyer informs the participants that the Temple Gastroenterology department is performing a health survey and gives them a phone number to call if they are interested. This phone is in a locked lab run by the PI. As compensation for their time they will receive $25. Only one subject per household is eligible and interviews can be completed at the hospital or in the participant's home. Only those individuals willing to be contacted in future years for follow-up will be enrolled. Subjects must show an identification verifying that their home address is in the zip code (usually a driver's license).

The overall survey consists of several standardized questionnaires which have been organized into a logical, easy to complete, comprehensive unit. Patients will complete the survey on a laptop which contains all the questions in an easy to read and follow Microsoft Access database file. Essentially no computer skills are needed to complete it except for the use of a mouse. A member of the research team will sit in the room to help the subject if there are questions. This survey is password secured such that when the subject completes the survey they cannot access the responses of other subjects. Answering the last question automatically closes the file.

The individual questionnaires making up the overall survey are included in this packet. Initial questions ask the subject their name, address, contact phone numbers and demographic questions such as income and education level. Subsequent questions are the complete set of questions from standardized questionnaires such as AUDIT for alcohol use assessment. The cornerstones of the survey are the 17 question survey on GERD which covers all components of the Montreal classification, and the 65 questions which make up the Rome III functional bowel disease questionnaire. We estimate it will take participants 30-60 minutes to complete depending on age and educational level.

Risks.

The only potential risk is related to confidentiality. Sensitive personal information is assessed using the survey. Several levels of subject protection will be employed. These include use of a password protected file for database collection on a computer which is password protected when turned off. The computer will be kept in a locked office in the hospital. The phone used to interact with subjects is in lab #7 of the Parkinson Pavilion, 10th floor.

There are no interventions to be performed for this study. There will be, for example, no blood draws. Future studies may recruit individuals from this database for invasive diagnostic testing and further data collection but those will be covered under future IRB submissions.

Benefits

Subjects who participate in the study will develop a greater insight into the possible causes of their medical problem. In a relaxed environment will they have the opportunity to talk with a board-certified gastroenterologist about their health. They will be provided with accurate information and will be encouraged to engage the health care system by communicating with their primary care physician. The African American community as a whole will benefit tremendously as their health status within the US is presented in peer-reviewed literature. This has the potential to shape public policy. Future studies under separate IRB protocols may provide benefit to them such as free testing for potentially serious GI diseases.

Data Collection and Statistics

We will recruit a minimum of 100 African Americans from each quadrant of the zip code 19140 with the total adding to 450.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* self-described African American or Caucasian
* lived in zip code for > 3 years

Exclusion Criteria:

* newly arrived to zip code
* unable to provide proof of address
* unwilling to come to temple to complete interview

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult individuals (age 18-80)residing in the 19140 zip code area will be eligible for participation. We will interview 750 African American residents and 250 self-described Caucasian residents.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2010-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank K Friedenberg, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | African Americans
Started | 450
Completed | 450
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 450 African Americans living around Temple Hospital
Arm/Group | African Americans
Number analyzed (Participants) | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272
  Male | 178
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 450
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 450

OUTCOME MEASURES:

1. Primary Outcome: Epidemiologic Factors Associated With Prevalent Reflux Disease.
Description: Patients will complete a series of standardized questionnaires to determine the prevalence of reflux disease and risk factors for its development. We will query diet, depression, drug, tobacco, and alcohol use as well as a variety of other factors. We will study 450 African Americans living in North Philadelphia.
Time Frame: Two years
Population: Patients successfully identified from targeted area.
Measure: Number (95% Confidence Interval); unit: percentage of participants with GERD
Arm/Group | African Americans
Number analyzed (Participants) | 450
percentage of participants with GERD | 17.6 [16.4 to 18.8]

ADVERSE EVENTS:
Arm/Group | African Americans
Serious Adverse Events (participants affected / at risk) | 0/450
Other Adverse Events (participants affected / at risk) | 0/450

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No